CLINICAL TRIAL: NCT04514666
Title: Exhaled Volatile Organic Compounds as Potential Predictive Biomarkers of Chronic Kidney and Liver Rejection After Transplants
Brief Title: VOCs in Kidney and Liver Transplants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Societa Italiana di Chirurgia ColoRettale (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38/2020
Record Dates: First submitted 2020-08-12; First posted 2020-08-17 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Liver Transplant Rejection; Kidney Transplant; Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver/kidney transplant (Experimental): The breath of patients undergoing liver or kidney transplant will be sampled and analysed
  Interventions: Other: Breath analysis

INTERVENTIONS:
Other: Breath analysis — The breath of patients undergoing liver or kidney transplant will be sampled and volatile organic compounds will be identified

SUMMARY:
Kidney and liver trasplants represent very challenging lifesaving and effective surgical procedures for patients with end-stage kidney and/or liver disease.

Chronic rejection may occur in 3 to 17% livers transplants and in 20 to 40% kidney transplants.

While acute rejection is clearly detected due to the clinical features and laboratory tools, the early identification of chronic rejection is still challenging since the clinical features are often silents and laboratory tests become suggestive when the damage due to the rejection is almost irreversible.

Considering the recent application of the breathomic to liver and kidney disease and the difficulty in the early detection of chronic rejection after liver and kidney transplants, the analysis of the exhaled VOCs pattern could help early detection of chronic rejection allowing a prompt medical treatment.

DETAILED DESCRIPTION:
Kidney and liver trasplants represent very challenging lifesaving and effective surgical procedures for patients with end-stage kidney and/or liver disease.

Nowadays the short and long term success rate of kidney and liver trasplants is pretty hight. Nevertheless, transplant rejection remains one of the biggest limitations with a strong impact on patients survival.

Usually acute rejection occurs within 3 months after the transplant and is the most common cause of transplant failure and the most common indication for re-transplantation .

Chronic rejection may occur in 3 to 17% livers transplants and in 20 to 40% kidney transplants.

While acute rejection is clearly detected due to the clinical features and laboratory tools, the early identification of chronic rejection is still challenging since the clinical features are often silents and laboratory tests become suggestive when the damage due to the rejection is almost irreversible.

Chronic renal transplant rejection is the result of a gradual decrease in the kidney function that starts to become evident three months after surgery.

Kidney chronic rejection is, by definition, immune-mediated and generally divides into chronic active antibody-mediated rejection and chronic active T cell-mediated rejection.

Transplant vasculopathy is the single most important feature of chronic renal transplant rejection and it is the direct consequence of an immune reaction that activates a cytokines cascade with a tissue fibrosis and chronic rejection.

Hypertension and proteinuria are the most important features of declining renal function.

Laboratory tests such as serum creatinine and estimated glomerular filtration rate (eGFR)ccan help to early identify kidney allograft dysfunction. The eGFR is suggested to be a more accurate indicator and predictor of graft function and long term graft loss.

However, a biopsy is mandatory for diagnosing chronic renal transplant rejection. C4d complement fragment deposition in the peritubular capillaries represents the marker for antibody-mediated tissue injury.

Although the incidence of acute and chronic rejection has declined with improvement of immunosuppression regimens, chronic rejection may lead to re-transplant or death.

Chronic liver allograft rejection usually occurs more than 2 months after transplantation and most frequently develops after an unresolved or multiple episodes of acute rejection or indolently over a period of months to years, with few or no clinically apparent acute cellular rejection episodes.

Chronic rejection characterized primarily by fibrointimal hyperplasia of arteries, or obliterative arteriopathy, interstitial fibrosis and atrophy of parenchymal elements.

Often the only reliable early indicator of chronic rejection is persistent and preferential elevation of γ-glutamyl transpeptidase and alkaline phosphatase, which is related to bile duct damage. In most of cases the only clinical sign is jaundice and it appears when allograft dysfunction becomes. Biliary sludging or appearance of biliary strictures, hepatic infarcts, and finally loss of hepatic synthetic function, which can manifest as coagulopathy, malnutrition, and hepatosplenomegaly are late findings presaging allograft failure. Biopsy is mandatory to assess the liver damage.

Breath analysis (Breathomics) is applied widely nowadays in clinical setting in order to identify and evaluate exhaled molecular volatile compounds as expression of a metabolic derangement of the organism including chronic diseases and cancer disease.

A novel approach, a breath test based on the metabolomic evaluation of the volatile organic compounds (VOCs) in the exhaled breath, has recently been developed by our group to identify patients with Colorectal cancer, showing good reliability and compliance.

VOCs analysis has also been demonstrated to find an application in the diagnosis of chronic liver and kidney disease with high sensitivity and specificity.

Considering the recent application of the breathomic to liver and kidney disease and the difficulty in the early detection of chronic rejection after liver and kidney transplants, the analysis of the exhaled VOCs pattern could help early detection of chronic rejection allowing a prompt medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Both sex
* Patients eligible for liver or kidney transplant
* Written informed consent

Exclusion Criteria:

* Acute liver failure
* Acute liver and kidney rejection
* HCC
* Re-transplant
* Pregnancy
* IBD
* Any psychiatric disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-02 (Estimated); Primary Completion 2022-10-02 (Estimated); Study Completion 2023-03-02 (Estimated)

PRIMARY OUTCOMES:
Volatile organic compounds in end stage liver disease | 30 days
  to evaluate the pattern of volatile organic compounds in patients elegible for liver transplant
Volatile organic compounds in end stage kidney disease | 30 days
  to evaluate the pattern of volatile organic compounds in patients elegible for kidney transplant
Volatile organic compounds after liver transplant | 1 year
  to evaluate the pattern of volatile organic compounds able to identify the onset of chronic failure/rejection after liver transplants
Volatile organic compounds after liver transplant | 1 year
  to evaluate the pattern of volatile organic compounds able to identify the onset of chronic failure/rejection after kidney transplants

CONTACTS AND LOCATIONS:
Overall Officials: Arcangelo Picciariello, MD, Principal Investigator — Societa Italiana di Chirurgia ColoRettale
Locations (1):
- Dept of Emergency and Organ transplantation, Bari, Italy

IPD SHARING:
Plan to Share IPD: Undecided